CLINICAL TRIAL: NCT04842526
Title: Efficacy and Safety of Anlotinib, Irinotecan and Temozolomide in the Treatment of Refractory or Recurrent Neuroblastoma in Children: an Open, Single Arm, Single Center, Phase II Clinical Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Qiang Zhao1
Record Dates: First submitted 2021-03-29; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-02

CONDITIONS: Refractory or Recurrent Neuroblastoma in Children
MeSH Terms: interventions — anlotinib; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib and irinotecan combined with temozolomide (Experimental)
  Interventions: Drug: Anlotinib and irinotecan combined with temozolomide

INTERVENTIONS:
Drug: Anlotinib and irinotecan combined with temozolomide — Anlotinib, 7mg/m2, PO, was given for 14 days and stopped for 7 days; Irinotecan, 50mg/m2, D1-5, IV; Temozolomide, 100mg/m2, d1-5, PO; Three weeks is a cycle.

SUMMARY:
Neuroblastoma is an embryonal tumor originated from primitive neural crest cells. It is the most common extracranial solid tumor in children. It is characterized by abundant blood vessels, rapid growth and early metastasis.With the gradual improvement of diagnosis and treatment technology, the survival rate of children with Neuroblastoma in China has been increasing year by year, but the Overall Survival is still lower than that in European and American countries, so new and efficient treatment methods are urgently needed in clinical practice.Anti-angiogenesis target therapy is an important component of the malignant tumor treatment, hydrochloric acid for Anlotinib has the anti-tumor angiogenesis and suppress tumor growth, Anlotinib currently in thyroid carcinoma, esophageal cancer, liver cancer, colorectal cancer, soft nest, cervical cancer, soft tissue sarcoma and so on the many kinds of cancer are conducting clinical trials, but in neuroblastoma application has not been reported.The purpose of this study was to explore the therapeutic effect and mechanism of Anlotinib and irinotecan combined with temozolomide in the treatment of refractory or recurrent Neuroblastoma in children.Neuroblastoma is an embryonal tumor originated from primitive neural crest cells. It is the most common extracranial solid tumor in children. It is characterized by abundant blood vessels, rapid growth and early metastasis.It accounts for 8%-10% of all malignant tumors in children, with an annual incidence of 0.3-5.5/100,000.The prognosis of Neuroblastoma was closely related to age at diagnosis, clinical stage, tumor pathological type, N-myc gene copy number and DNA index.According to the above five indicators, the Children's Oncology Group divided NB into low, medium and high risk groups.According to the 2013 Children's Oncology Group data, the current 5-year Overall Survival of low - and moderate-risk Neuroblastoma patients was 90%, while the Overall Survival of high-risk patients was only 50%.The current treatment of Neuroblastoma is a multidisciplinary combination of surgery, chemoradiotherapy and autologous stem cell transplantation.With the gradual improvement of diagnosis and treatment technology, the survival rate of children with NB in China has been increasing year by year, but the Overall Survival is still lower than that in European and American countries, so new and efficient treatment methods are urgently needed in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent was signed before admission;
2. Under 21 years old, both male and female;
3. Patients with distant metastasis or locally advanced neuroblastoma judged by the researchers to be unsuitable for surgical treatment;
4. According to RECIST v1.1, at least one measurable lesion was judged by CT or MRI;
5. Patients who have used at least one chemotherapy regimen (including anthracycline) for treatment and are evaluated as disease progression or intolerable according to RECIST 1.1;
6. PS score: 0-1 (for amputees, it can be relaxed to 2); the expected survival time is more than 12 weeks;
7. At least 2 weeks after the last biotherapy and 3 weeks after the last chemotherapy;
8. All acute toxicity reactions caused by previous anti-tumor therapy or surgery were alleviated to 0-1 level before the screening period (according to NCI CTCAE 5.0) or to the level specified by the inclusion / exclusion criteria (except for the toxicity of alopecia, etc., which was considered by the researchers to have no safety risk to the subjects).
9. Adequate organ and bone marrow functions are defined as follows:

   routine blood test

   Neutrophil count (ANC) ≥ 1000 / mm3 (1.0 × 109 / L);

   Platelet count (PLT) ≥ 70000 / mm3 (70 × 109 / L);

   Hemoglobin (HB) ≥ 7.5 g / dl (75 g / L);

   Blood biochemistry

   Serum creatinine (CR) ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance rate (cockroft Gault)

   Total bilirubin (TBIL) ≤ 1.5 × ULN;

   Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≤ 2.5 × ULN, liver metastasis subjects should be ≤ 5 × ULN;

   Coagulation function

   International normalized ratio (INR) ≤ 1.5, prothrombin time (PT) and activated partial thromboplastin

   （APTT）≤1.5×ULN；

   urinalysis

   Urinary protein < 2 +; if urinary protein ≥ 2 +, 24-hour urinary protein quantitative display protein must be ≤ 1g;

   Cardiac function

   Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ lower limit of normal value (50%)
10. All women of childbearing age should be given adequate contraceptive treatment before and after 7 weeks of pregnancy.
11. The subjects voluntarily or their legal guardians agreed to join the study, with good compliance and follow-up of safety and survival.

Exclusion Criteria:

1. Received the following treatment within 3 weeks before treatment:

   Radiotherapy, surgery, chemotherapy and molecular targeted therapy for tumors;

   Other clinical research drugs;

   Live attenuated vaccine.
2. Patients who had received anti angiogenic targeted drugs in the past 3 months, such as apatinib, pazoparib, sunitinib, sorafenib, bevacizumab, imatinib, clotriminib, famitinib, anlotinib, repaglinide, endostatin, etc.
3. Patients who have previously received irinotecan or combined with temozolomide for progression.
4. Surgery and / or radiotherapy for solid tumors were planned during the study period (regardless of < 5% of bone marrow areas).
5. Long term unhealed wounds, ulcers or fractures, major surgery 28 days before enrollment or minor surgery 7 days before enrollment, known bleeding tendency, history of thrombosis 3 months before enrollment, cerebrovascular events, abdominal fistula, gastrointestinal perforation, abdominal abscess 6 months before enrollment, known brain metastasis.
6. Severe infection (e.g. intravenous antibiotics, antifungal or antiviral drugs) occurred within 1 week before treatment, or fever of unknown origin > 38.5 ° C occurred during screening / before the first administration.
7. Hypertension could not be well controlled by antihypertensive drugs (infants > 100 / 60mmhg, preschool children (< 6 years old) > 110 / 70mmhg, school-age children (6-12 years old) > 120 / 80mmHg, adolescence and adults (> 18 years old) > 140 / 90mmHg).
8. There were significant clinical bleeding symptoms or clear bleeding tendency within 3 months before treatment, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood + + and above, vasculitis, etc.; or arteriovenous thrombosis events within 6 months before treatment, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism Long term anticoagulant therapy with warfarin or heparin or long-term antiplatelet therapy (aspirin ≥ 300 mg / day or clopidogrel ≥ 75 mg / day) is needed.
9. There were active heart diseases, including myocardial infarction, severe / unstable angina pectoris, etc. within 6 months before treatment. The left ventricular ejection fraction (LVEF) was less than 50% and the arrhythmias were poorly controlled (including QTCF interval > 450 ms in male and > 470 MS in female).
10. Any other malignant tumor was diagnosed within 3 years before treatment.
11. Known to be allergic to the study drug or any of its excipients.
12. Human immunodeficiency virus (HIV) infection, active hepatitis B (HBsAg positive and HBV DNA ≥ 500 IU / ml), hepatitis C (HCV antibody positive and HCV-RNA higher than the detection limit of the analytical method).
13. The patients with huge tumor, easy to burst and bleeding, tumor regression, easy to lead to bleeding and other high-risk patients.
14. According to the judgment of the researcher, there are concomitant diseases (such as poorly controlled hypertension, severe diabetes, neurological or mental diseases, etc.) or any other conditions that seriously endanger the safety of the subject, may confuse the results of the study, or affect the completion of the study.

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-04-12 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | up to six months
  Randomization began until the first tumor progression or time of death